CLINICAL TRIAL: NCT00845728
Title: A Phase IIIb Multicenter, 52 Week Treatment, Randomized, Blinded, Double Dummy, Parallel Group Efficacy Study Comparing the Effect of Inhaled Indacaterol 150 µg o.d. vs Inhaled Tiotropium 18 µg o.d. on Lung Function, Rate of Exacerbations and Related Outcomes in Patients With COPD
Brief Title: Exacerbation Study
Acronym: INVIGORATE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQAB149B2348; 2008-007944-33
Record Dates: First submitted 2009-02-15; First posted 2009-02-18 (Estimated); Results first posted 2013-11-19 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Indacaterol; Tiotropium; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Indacaterol (Experimental): Indacaterol 150 µg o.d. delivered via single-dose dry powder inhaler (SDDPI)
  Interventions: Drug: Indacaterol 150 µg
- Tiotropium (Active Comparator): Tiotropium 18 µg o.d. delivered via the handihaler®
  Interventions: Drug: Tiotropium

INTERVENTIONS:
Drug: Indacaterol 150 µg — Indacaterol 150 µg o.d. delivered via SDDPI
  Arms: Indacaterol
Drug: Tiotropium — Tiotropium 18 µg o.d. delivered via handihaler®
  Arms: Tiotropium

SUMMARY:
This study compares indacaterol with tiotropium in terms of bronchodilation over 52 weeks

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults aged ≥40 years, who have signed an Informed Consent form prior to initiation of any study-related procedure
* Patients diagnosed with COPD at age 40 and over and with a current diagnosis of severe COPD and including:

  1. Smoking history of at least 10 pack years, both current and ex-smokers are eligible
  2. A documented history of at least 1 moderate or severe exacerbation in the previous 12 months

Exclusion Criteria:

* Patients who have received systemic corticosteroids and/or antibiotics for a COPD exacerbation in the 6 weeks prior to screening or during the run-in period
* Patients who have had a respiratory tract infection within 6 weeks prior to screening
* Patients with concomitant pulmonary disease
* Patients with a history of asthma
* Patients with diabetes Type I or uncontrolled diabetes Type II
* Any patient with lung cancer or a history of lung cancer
* Patients with a history of certain cardiovascular comorbid conditions

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3439 (Actual)
Dates: Start 2009-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (353):
- Argentina (7):
  - Novartis Investigative Site, Buenos Aires, Buenos Aires
  - Novartis Investigative Site, Capital Federal, Buenos Aires
  - Novartis Investigative Site, Mar del Plata, Buenos Aires
  - Novartis Investigative Site, Pilar, Buenos Aires
  - Novartis Investigative Site, Mendoza, Mendoza Province
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, San Miguel de Tucumán, Tucumán Province
- Australia (7):
  - Novartis Investigative Site, Bankstown, New South Wales
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, Daw Park, South Australia
  - Novartis Investigative Site, Heidelberg, Victoria
  - Novartis Investigative Site, Parkville, Victoria
  - Novartis Investigative Site, Nedlands, Western Australia
  - Novartis Investigative Site, Tauranga, New Zealand
- Austria (7):
  - Novartis Investigative Site, Feldbach, Austria
  - Novartis Investigative Site, Gänserndorf, Austria
  - Novartis Investigative Site, Grieskirchen, Austria
  - Novartis Investigative Site, Hallein, Austria
  - Novartis Investigative Site, Linz, Austria
  - Novartis Investigative Site, Perg, Austria
  - Novartis Investigative Site, Zwettl Stadt, Austria
- Belgium (22):
  - Novartis Investigative Site, Framerie, Belgium
  - Novartis Investigative Site, Geraardsbergen, Belgium
  - Novartis Investigative Site, Gilly, Belgium
  - Novartis Investigative Site, Malmedy, Belgium
  - Novartis Investigative Site, Menen, Belgium
  - Novartis Investigative Site, Aalst
  - Novartis Investigative Site, Antwerp
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Duffel
  - Novartis Investigative Site, Eupen
  - Novartis Investigative Site, Godinne
  - Novartis Investigative Site, Gozée
  - Novartis Investigative Site, Herentals
  - Novartis Investigative Site, Jambes
  - Novartis Investigative Site, Jette
  - Novartis Investigative Site, Kortrijk
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
  - Novartis Investigative Site, Montigny-le-Tilleul
  - Novartis Investigative Site, Namur
  - Novartis Investigative Site, Ostend
  - Novartis Investigative Site, Turnhout
- Brazil (6):
  - Novartis Investigative Site, Goiânia, Goiás
  - Novartis Investigative Site, Juiz de Fora, Minas Gerais
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Caxias do Sul, Rio Grande do Sul
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, São Paulo, São Paulo
- Canada (14):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Kelowna, British Columbia
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Winnipeg, Manitoba
  - Novartis Investigative Site, Moncton, New Brunswick
  - Novartis Investigative Site, Burlington, Ontario
  - Novartis Investigative Site, Mississauga, Ontario
  - Novartis Investigative Site, Newmarket, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Sainte-Foy, Quebec
  - Novartis Investigative Site, Sherbrooke, Quebec
- China (8):
  - Novartis Investigative Site, Shijiazhuang, Hebei
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Shengyang, Liaoning
  - Novartis Investigative Site, Xi’an, Shanxi
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Chongqing
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Shenyang
- Colombia (3):
  - Novartis Investigative Site, Barranquilla
  - Novartis Investigative Site, Bogotá
  - Novartis Investigative Site, Medellín
- Costa Rica (2):
  - Novartis Investigative Site, San Francisco de Asís, Costa Rica
  - Novartis Investigative Site, San José, Costa Rica
- Czechia (17):
  - Novartis Investigative Site, Beroun, Czech Republic
  - Novartis Investigative Site, Cvikov, Czech Republic
  - Novartis Investigative Site, České Budějovice, Czech Republic
  - Novartis Investigative Site, Český Krumlov, Czech Republic
  - Novartis Investigative Site, Karlovy Vary, Czech Republic
  - Novartis Investigative Site, Kuřim, Czech Republic
  - Novartis Investigative Site, Ostrava, Czech Republic
  - Novartis Investigative Site, Ostrava - Hrabuvka, Czech Republic
  - Novartis Investigative Site, Prague, Czech Republic
  - Novartis Investigative Site, Přerov, Czech Republic
  - Novartis Investigative Site, Rokycany, Czech Republic
  - Novartis Investigative Site, Rudná, Czech Republic
  - Novartis Investigative Site, Strakonice, Czech Republic
  - Novartis Investigative Site, Teplice, Czech Republic
  - Novartis Investigative Site, Žatec, Czech Republic
  - Novartis Investigative Site, Kyjov, CZE
  - Novartis Investigative Site, Nový Jičín
- Denmark (7):
  - Novartis Investigative Site, Aalborg, Denmark
  - Novartis Investigative Site, Elsinore, Denmark
  - Novartis Investigative Site, Hellerup, Denmark
  - Novartis Investigative Site, Hvidovre, Denmark
  - Novartis Investigative Site, Aarhus
  - Novartis Investigative Site, Copenhagen NV
  - Novartis Investigative Site, Odense C
- Estonia (3):
  - Novartis Investigative Site, Tartu, Estonia
  - Novartis Investigative Site, Rakvere
  - Novartis Investigative Site, Tallinn
- Finland (7):
  - Novartis Investigative Site, Helsinki, Finland
  - Novartis Investigative Site, Jyväskylä, Finland
  - Novartis Investigative Site, Turku, Finland
  - Novartis Investigative Site, HUS
  - Novartis Investigative Site, Pori
  - Novartis Investigative Site, Porvoo
  - Novartis Investigative Site, Tampere
- France (14):
  - Novartis Investigative Site, Beuvry, France
  - Novartis Investigative Site, Bourges, France
  - Novartis Investigative Site, Ferolles-Attily, France
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Ollioules
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Perpignan
  - Novartis Investigative Site, Pessac
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Saint-Michel-sur-Orge
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
- Germany (29):
  - Novartis Investigative Site, Berlin, Germany
  - Novartis Investigative Site, Leipzig, Germany
  - Novartis Investigative Site, Mainz, Germany
  - Novartis Investigative Site, Marburg, Germany
  - Novartis Investigative Site, München, Germany
  - Novartis Investigative Site, Teterow, Germany
  - Novartis Investigative Site, Bad Wörishofen
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Borstel
  - Novartis Investigative Site, Dachau
  - Novartis Investigative Site, Euskirchen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Fürstenwalde
  - Novartis Investigative Site, Güstrow
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hoyerswerda
  - Novartis Investigative Site, Landsberg
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Neu-Ulm
  - Novartis Investigative Site, Neumünster
  - Novartis Investigative Site, Neuss
  - Novartis Investigative Site, Oranienburg
  - Novartis Investigative Site, Radebeul
  - Novartis Investigative Site, Ratingen
  - Novartis Investigative Site, Rüdersdorf
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Wedel
  - Novartis Investigative Site, Witten
- Hungary (10):
  - Novartis Investigative Site, Cegléd, Hungary
  - Novartis Investigative Site, Debrecen, Hungary
  - Novartis Investigative Site, Szarvas, Hungary
  - Novartis Investigative Site, Tatabánya, Hungary
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Deszk
  - Novartis Investigative Site, Mosonmagyaróvár
  - Novartis Investigative Site, Nyíregyháza
  - Novartis Investigative Site, Sopron
  - Novartis Investigative Site, Törökbálint
- Novartis Investigative Site, Reykjavik, Iceland
- India (16):
  - Novartis Investigative Site, Hyderabad, Andhra Pradesh
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Ahmedabad, Gujrat-India
  - Novartis Investigative Site, Nagpur - Maharashtra, India
  - Novartis Investigative Site, Nagpur - Maharastra, India
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Mangalore, Karnataka
  - Novartis Investigative Site, Calicut, Kerala
  - Novartis Investigative Site, Trivandrum, Kerala
  - Novartis Investigative Site, Indore, Madhya Pradesh
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Noida, New Delhi
  - Novartis Investigative Site, Jaipur, Rajasthan
  - Novartis Investigative Site, Coimbatore, Tamil Nadu
  - Novartis Investigative Site, Vellore, Tamil Nadu
  - Novartis Investigative Site, Panjim
- Israel (5):
  - Novartis Investigative Site, Ashkelon
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Rehovot
  - Novartis Investigative Site, Tel Aviv
- Italy (24):
  - Novartis Investigative Site, Acquaviva delle Fonti, BA
  - Novartis Investigative Site, Bari, BA
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Catanzaro, CZ
  - Novartis Investigative Site, Cona, FE
  - Novartis Investigative Site, Cassino, FR
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Pisa, Italy
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Pordenone, PN
  - Novartis Investigative Site, Prato, PO
  - Novartis Investigative Site, Parma, PR
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Cava de' Tirreni, SA
  - Novartis Investigative Site, Siena, SI
  - Novartis Investigative Site, Teramo, TE
  - Novartis Investigative Site, Orbassano, TO
  - Novartis Investigative Site, Trieste, TS
  - Novartis Investigative Site, Cuasso al Monte, VA
  - Novartis Investigative Site, Verona, VR
  - Novartis Investigative Site, Napoli
- Latvia (2):
  - Novartis Investigative Site, Riga, LV
  - Novartis Investigative Site, Riga
- Lithuania (5):
  - Novartis Investigative Site, Kaunas
  - Novartis Investigative Site, Klaipėda
  - Novartis Investigative Site, Šiauliai
  - Novartis Investigative Site, Utena
  - Novartis Investigative Site, Vilnius
- Mexico (4):
  - Novartis Investigative Site, Pachuca, Hidalgo
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, Monterrey, Nuevo León
  - Novartis Investigative Site, San Luis Potosí City, San Luis Potosí
- Netherlands (7):
  - Novartis Investigative Site, Almelo, Netherlands
  - Novartis Investigative Site, Breda, Netherlands
  - Novartis Investigative Site, Enschede, Netherlands
  - Novartis Investigative Site, Eindhoven
  - Novartis Investigative Site, Rotterdam
  - Novartis Investigative Site, Sneek
  - Novartis Investigative Site, Zwolle
- Peru (9):
  - Novartis Investigative Site, Jesus Maria, Lima region
  - Novartis Investigative Site, La Victoria, Lima region
  - Novartis Investigative Site, Lima Cercado, Lima region
  - Novartis Investigative Site, Miraflores, Lima region
  - Novartis Investigative Site, San Borja, Lima region
  - Novartis Investigative Site, San Isidro, Lima region
  - Novartis Investigative Site, San Martín de Porres, Lima region
  - Novartis Investigative Site, San Miguel, Lima region
  - Novartis Investigative Site, Santiago de Surco, Lima region
- Philippines (3):
  - Novartis Investigative Site, Quezon City, National Capital Region
  - Novartis Investigative Site, Quezon City, Philippines
  - Novartis Investigative Site, Quezon City
- Poland (5):
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Katowice
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
- Portugal (4):
  - Novartis Investigative Site, Amadora
  - Novartis Investigative Site, Coimbra
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Porto
- Romania (6):
  - Novartis Investigative Site, Bucharest, District 3
  - Novartis Investigative Site, Brasov, Jud. Brasov
  - Novartis Investigative Site, Constanța, Jud. Constanta
  - Novartis Investigative Site, Iași, Jud. Iasi
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Cluj-Napoca
- Russia (7):
  - Novartis Investigative Site, Kazan', Tatarstan Republic
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Samara
  - Novartis Investigative Site, Yekaterinburg
- Slovakia (8):
  - Novartis Investigative Site, Bratislava, Slovak Republic
  - Novartis Investigative Site, Košice, Slovak Republic
  - Novartis Investigative Site, Spišská Nová Ves, Slovak Republic
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Lučenec
  - Novartis Investigative Site, Nové Zámky
  - Novartis Investigative Site, Poprad
- South Africa (3):
  - Novartis Investigative Site, Durban, South Africa
  - Novartis Investigative Site, Bloemfontein
  - Novartis Investigative Site, Cape Town
- Spain (23):
  - Novartis Investigative Site, Jerez de la Frontera, Andalusia
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Sanlúcar de Barrameda, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Valladolid, Castille and León
  - Novartis Investigative Site, Illescas, Castille-La Mancha
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Salt, Catalonia
  - Novartis Investigative Site, Sant Boi de Llobregat, Catalonia
  - Novartis Investigative Site, Terrassa, Catalonia
  - Novartis Investigative Site, Vic, Catalonia
  - Novartis Investigative Site, Cáceres, Extremadura
  - Novartis Investigative Site, Mérida, Extremadura
  - Novartis Investigative Site, Plasencia, Extremadura
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Lugo, Galicia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Madrid, Madrid
  - Novartis Investigative Site, Pozuelo de Alarcón, Madrid
  - Novartis Investigative Site, Gijón, Principality of Asturias
  - Novartis Investigative Site, Alicante, Valencia
  - Novartis Investigative Site, Alzira, Valencia
  - Novartis Investigative Site, Requena, Valencia
- Sweden (7):
  - Novartis Investigative Site, Skellefteå, Sweden
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Luleå
  - Novartis Investigative Site, Lund
  - Novartis Investigative Site, Malmo
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Sundsvall
- Switzerland (8):
  - Novartis Investigative Site, Faltigberg-Wald, Canton of Zurich
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Crans-Montana
  - Novartis Investigative Site, Lausanne
  - Novartis Investigative Site, Sankt Gallen
  - Novartis Investigative Site, Thun
  - Novartis Investigative Site, Winterthur
  - Novartis Investigative Site, Zurich
- Taiwan (4):
  - Novartis Investigative Site, Taichung, Taiwan
  - Novartis Investigative Site, Taipei, Taiwan
  - Novartis Investigative Site, Taipei County, Taiwan
  - Novartis Investigative Site, Taipei
- Thailand (4):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
  - Novartis Investigative Site, Khon Kaen
  - Novartis Investigative Site, Songkhla
- Turkey (Türkiye) (14):
  - Novartis Investigative Site, Ankara, Turkey
  - Novartis Investigative Site, Isparta, Turkey
  - Novartis Investigative Site, Kahramanmaraş, Turkey
  - Novartis Investigative Site, Çanakkale
  - Novartis Investigative Site, Diskapi / Ankara
  - Novartis Investigative Site, Emek / Ankara
  - Novartis Investigative Site, Gaziantep
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Kecioren / Ankara
  - Novartis Investigative Site, Kozlu / Zonguldak
  - Novartis Investigative Site, Malatya
  - Novartis Investigative Site, Mersin
  - Novartis Investigative Site, Yenisehir/Izmir
- United Kingdom (18):
  - Novartis Investigative Site, Swansea, England
  - Novartis Investigative Site, Newcastle upon Tyne, Newcastle
  - Novartis Investigative Site, Ash Vale, Surrey
  - Novartis Investigative Site, Cambridge, United KIngdom
  - Novartis Investigative Site, Watford, United Kingdom
  - Novartis Investigative Site, Crawley, West Sussex
  - Novartis Investigative Site, Belfast
  - Novartis Investigative Site, Bexhill-on-Sea
  - Novartis Investigative Site, Bradford
  - Novartis Investigative Site, Bristol
  - Novartis Investigative Site, Lancashire
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Newport
  - Novartis Investigative Site, Stockport
  - Novartis Investigative Site, Surrey
  - Novartis Investigative Site, Warminster
  - Novartis Investigative Site, Windsor
- Venezuela (3):
  - Novartis Investigative Site, Valencia, Carabobo
  - Novartis Investigative Site, Barquisimeto, Lara
  - Novartis Investigative Site, Maracaibo, Zulia

REFERENCES:
- [Derived] Decramer ML, Chapman KR, Dahl R, Frith P, Devouassoux G, Fritscher C, Cameron R, Shoaib M, Lawrence D, Young D, McBryan D; INVIGORATE investigators. Once-daily indacaterol versus tiotropium for patients with severe chronic obstructive pulmonary disease (INVIGORATE): a randomised, blinded, parallel-group study. Lancet Respir Med. 2013 Sep;1(7):524-33. doi: 10.1016/S2213-2600(13)70158-9. Epub 2013 Aug 21. PMID 24461613

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 3,444 patients were randomized, but only 3,439 received treatment as 5 patients were mis-randomized.
Groups:
- Indacaterol: Indacaterol 150 μg o.d., delivered via SDDPI o.d. plus placebo to tiotropium o.d.
  delivered via the manufacturer's proprietary inhalation device (Handihaler®)
- Tiotropium: Tiotropium 18 μg o.d. delivered via the manufacturer's proprietary inhalation device (Handihaler®) plus placebo to indacaterol o.d. delivered via SDDPI
Period: Overall Study
Arm/Group | Indacaterol | Tiotropium
Started | 1723 | 1721
Exposed | 1721 | 1718
Completed | 1337 | 1379
Not Completed | 386 | 342
Not completed — Abnormal laboratory value (s) | 2 | 2
Not completed — Patient's inability to use the device | 4 | 6
Not completed — Abnormal test procedure result (s) | 7 | 2
Not completed — Lost to Follow-up | 22 | 13
Not completed — Death | 24 | 26
Not completed — Administrative Problems | 34 | 26
Not completed — Protocol Violation | 36 | 24
Not completed — Lack of Efficacy | 51 | 39
Not completed — Adverse Event | 101 | 96
Not completed — Withdrawal by Subject | 105 | 108

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Indacaterol | Tiotropium | Total
Number analyzed (Participants) | 1721 | 1718 | 3439
Age, Customized [Number; unit: Participants]
  <65 years | 929 | 909 | 1838
  ≥ 65 years | 792 | 809 | 1601
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 377 | 405 | 782
  Male | 1344 | 1313 | 2657

OUTCOME MEASURES:

1. Primary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1).
Description: The primary objective of the study was to demonstrate the non-inferiority of indacaterol vs. tiotropium with respect to 24 hour post dose (trough) FEV1 after 12 weeks of treatment in patients with severe COPD. Trough FEV1 was defined as the average of the 23 hours 10 min and the 23 hours 45 min post dose values. Trough FEV1 was analyzed using a mixed model for the PPS-S. The model contained treatment as a fixed effect with the baseline FEV1, FEV1 prior to inhalation and FEV1 15 min post-inhalation of salbutamol/albuterol (components of SABA reversibility at Visit 2), FEV1 prior to inhalation and FEV1 60 min post-inhalation of ipratropium (components of anti-cholinergic reversibility at Visit 3) as covariates. Smoking history (current or ex-smoker) was included as a factor in the model.
Time Frame: 12 weeks
Population: Per-Protocol Set for Spirometry (PPS-S) This set included Full Analysis Set (FAS) patients without any major protocol deviations or non-protocol deviation criteria that could affect the respective analysis of efficacy.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol | Tiotropium
Number analyzed (Participants) | 1450 | 1467
Liters | 1.134 (0.0008) | 1.145 (0.0008)

2. Secondary Outcome: Rate of COPD Exacerbations
Description: COPD exacerbations were defined as :Worsening of 2 or more major symptoms for at least 2 consecutive days: dyspnea; sputum volume; suputum purulence AND requiring treatment with systemic corticosteroids and/or antibiotics OR Worsening of any 1 major symptom together with any 1 of the following minor symptoms for at least 2 consecutive days: Sore throat; colds; fever without other cause; increased cough; increase wheeze AND requiring treatment with systemic glucocorticosteroids and/or antibiotics. The rate was analyzed using a linear model assuming a negative binomial distribution for the PPS-E. The time at risk for a patient was defined as the length of time the patient was in the study and the log(length of time in the study) was used as the offset variable in the model.
Time Frame: 52 weeks
Population: Per-Protocol Set for Exacerbations (PPS-E). This set included Full Analysis Set (FAS) patients without any major protocol deviations or non-protocol deviation criteria that could affect the respective analysis of efficacy.
Measure: Number; unit: Exacerbations per patient per year
Arm/Group | Indacaterol | Tiotropium
Number analyzed (Participants) | 1675 | 1675
Exacerbations per patient per year | 0.79 | 0.61

ADVERSE EVENTS:
Groups:
- IndIndacaterol: Indacaterol 150 μg o.d., delivered via SDDPI o.d. plus placebo to tiotropium o.d. delivered via the manufacturer's proprietary inhalation device (Handihaler®)
Arm/Group | IndIndacaterol | Tiotropium
Serious Adverse Events (participants affected / at risk) | 263/1721 | 255/1718
Other Adverse Events (participants affected / at risk) | 890/1721 | 793/1718
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IndIndacaterol (N=1721) | Tiotropium (N=1718)
Anaemia (Blood and lymphatic system disorders) | 0 | 3
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 3 | 2
Angina pectoris (Cardiac disorders) | 5 | 5
Angina unstable (Cardiac disorders) | 0 | 1
Aortic valve calcification (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 3 | 1
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 4
Atrial flutter (Cardiac disorders) | 2 | 1
Atrioventricular block (Cardiac disorders) | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Bundle branch block left (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 3 | 2
Cardiac failure (Cardiac disorders) | 3 | 5
Cardiac failure chronic (Cardiac disorders) | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 3 | 1
Cardio-respiratory arrest (Cardiac disorders) | 3 | 2
Cardiomegaly (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1
Cor pulmonale (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 3
Cyanosis (Cardiac disorders) | 0 | 1
Diastolic dysfunction (Cardiac disorders) | 1 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1
Left ventricular hypertrophy (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 4 | 8
Myocardial ischaemia (Cardiac disorders) | 6 | 4
Palpitations (Cardiac disorders) | 0 | 1
Right ventricular failure (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1
Supraventricular extrasystoles (Cardiac disorders) | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 1 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Goitre (Endocrine disorders) | 1 | 0
Angle closure glaucoma (Eye disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 1
Maculopathy (Eye disorders) | 0 | 1
Retinal vein occlusion (Eye disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Acute abdomen (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 3
Colonic polyp (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Diverticulum (Gastrointestinal disorders) | 1 | 0
Duodenal fistula (Gastrointestinal disorders) | 1 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 2
Enteritis (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 2
Gastritis (Gastrointestinal disorders) | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2
Haematemesis (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 3 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 3
Pancreatitis acute (Gastrointestinal disorders) | 0 | 2
Regurgitation (Gastrointestinal disorders) | 1 | 0
Sigmoiditis (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Cholangitis acute (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 1 | 2
Gallbladder fistula (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0
Appendicitis perforated (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 3 | 2
Bronchitis bacterial (Infections and infestations) | 1 | 1
Bronchopneumonia (Infections and infestations) | 2 | 3
Clostridial infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 2
Gastroenteritis (Infections and infestations) | 0 | 2
H1N1 influenza (Infections and infestations) | 1 | 0
Helicobacter infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 4
Influenza (Infections and infestations) | 4 | 2
Intervertebral discitis (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 4 | 4
Lower respiratory tract infection (Infections and infestations) | 28 | 18
Lower respiratory tract infection bacterial (Infections and infestations) | 4 | 2
Lower respiratory tract infection viral (Infections and infestations) | 0 | 1
Lung abscess (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 2
Meningitis (Infections and infestations) | 0 | 1
Meningitis viral (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 3 | 3
Oral candidiasis (Infections and infestations) | 0 | 1
Pneumococcal sepsis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 29 | 24
Pneumonia bacterial (Infections and infestations) | 1 | 2
Pneumonia pneumococcal (Infections and infestations) | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 1
Pseudomonas infection (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Respiratory tract infection bacterial (Infections and infestations) | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 2
Septic shock (Infections and infestations) | 1 | 3
Sinusitis (Infections and infestations) | 1 | 0
Testicular abscess (Infections and infestations) | 0 | 1
Tracheobronchitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 2
Upper respiratory tract infection bacterial (Infections and infestations) | 18 | 16
Urinary tract infection (Infections and infestations) | 1 | 2
Urosepsis (Infections and infestations) | 1 | 0
Viral sepsis (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 12 | 11
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 2
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 2
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 2
Penetrating abdominal trauma (Injury, poisoning and procedural complications) | 0 | 1
Post procedural fistula (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 2 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Traumatic shock (Injury, poisoning and procedural complications) | 0 | 1
Arteriogram coronary (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 1 | 0
Prostatic specific antigen increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Axillary mass (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Benign neoplasm of prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 5
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 | 0
Brain injury (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 2 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 1
Cerebral thrombosis (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 1
Coma (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Grand mal convulsion (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 0
Hypoglycaemic coma (Nervous system disorders) | 1 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 1
Intracranial aneurysm (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 2 | 0
Lacunar infarction (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 1
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Sensory loss (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 2 | 4
Vascular encephalopathy (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 2
Completed suicide (Psychiatric disorders) | 0 | 2
Confusional state (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 0 | 1
Bladder neck obstruction (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 2 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 3 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 3
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 147 | 121
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Aortic aneurysm (Vascular disorders) | 2 | 0
Aortic stenosis (Vascular disorders) | 2 | 0
Circulatory collapse (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 1
Hypertensive crisis (Vascular disorders) | 1 | 1
Hypertensive emergency (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Peripheral artery stenosis (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 0 | 1
Varicose vein (Vascular disorders) | 0 | 1
Chills (General disorders) | 1 | 0
Death (General disorders) | 1 | 1
Device dislocation (General disorders) | 1 | 0
Drug ineffective (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 4 | 1
Oedema due to cardiac disease (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 2 | 1
Pyrexia (General disorders) | 3 | 1
Soft tissue inflammation (General disorders) | 1 | 0
Sudden cardiac death (General disorders) | 0 | 1
Sudden death (General disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IndIndacaterol (N=1721) | Tiotropium (N=1718)
Diarrhoea (Gastrointestinal disorders) | 26 | 43
Bronchitis (Infections and infestations) | 39 | 34
Influenza (Infections and infestations) | 38 | 45
Lower respiratory tract infection (Infections and infestations) | 125 | 98
Nasopharyngitis (Infections and infestations) | 118 | 101
Upper respiratory tract infection (Infections and infestations) | 70 | 63
Upper respiratory tract infection bacterial (Infections and infestations) | 139 | 127
Urinary tract infection (Infections and infestations) | 31 | 26
Viral upper respiratory tract infection (Infections and infestations) | 91 | 65
Back pain (Musculoskeletal and connective tissue disorders) | 39 | 40
Headache (Nervous system disorders) | 53 | 49
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 668 | 591
Cough (Respiratory, thoracic and mediastinal disorders) | 107 | 56
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 56 | 50
Hypertension (Vascular disorders) | 63 | 48
Pyrexia (General disorders) | 19 | 26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are NOT employed by the organization sponsoring the study. Other disclosure agreement that restricts the right of the PI to discuss or publish trial results after the trial is completed.

The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial.